CLINICAL TRIAL: NCT07331558
Title: Effects of Multimodal Virtual Reality-based Rehabilitation on Dyspnea, Cardiorespiratory Fitness, Left Ventricular Ejection Fraction, and Quality of Life in CABG Phase II
Brief Title: Multimodal VR Rehabilitation for Cardiorespiratory Fitness in CABG Phase II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Amna Zafar
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: CABG
Keywords: multimodal treatment; virtual reality; telerehabilitation; education; Circuit Based Exercise; diet; psychological well-being
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Group A: Patients will engage in multimodal circuit training while simultaneously viewing nature scenes through VR in a clinical setting.
  Interventions: Other: multimodal circuit training while viewing nature scenes through VR in a clinical setting
- Group B (Experimental): Group B: Patients will be given multimodal circuit training in real -world clinical setting.
  Interventions: Other: multimodal circuit training in a real-world clinical setting
- Group C (Experimental): Group C: Patients will be given multimodal circuit training through telerehabilitation.
  Interventions: Other: multimodal circuit training through telerehabilitation

INTERVENTIONS:
Other: multimodal circuit training while viewing nature scenes through VR in a clinical setting — This will take place in a clinical setting where participants will also view the nature scenes through virtual reality (VR). The approach is multimodal, incorporating education through a booklet, physical activity via circuit training, nutritional counselling with a healthy diet prescription, and psychological well-being enhanced by behavioural cognitive therapy.
  Arms: Group A
Other: multimodal circuit training in a real-world clinical setting — This will take place in a real-world clinical setting. The approach is multimodal, incorporating education through a booklet, physical activity via circuit training, nutritional counselling with a healthy diet prescription, and psychological well-being enhanced by behavioural cognitive therapy.
  Arms: Group B
Other: multimodal circuit training through telerehabilitation — This will take place through Google Meetings. The approach is multimodal, incorporating education through a booklet, physical activity via circuit training, nutritional counselling with a healthy diet prescription, and psychological well-being enhanced by behavioural cognitive therapy.
  Arms: Group C

SUMMARY:
It will be a randomized clinical trial with a sample size of 66. A convenient sampling technique will be used to recruit the CABG phase II patients for the study. Then, they will be divided into three groups by block randomization. Weight-bearing Liuzijue Qigong will be given as a baseline treatment to all groups. In group A, patients will engage in multimodal circuit training while simultaneously viewing the nature scenes through VR in a clinical setting, in group B, patients will be given multimodal circuit training in a clinical setting while in group C, patients will be given multimodal circuit training through telerehabilitation. The dyspnea 12 Questionnaire will be used for measuring dyspnea, Cooper's 12-minute test will be used to assess cardiorespiratory fitness, echocardiography will be used to assess Left ventricular ejection fraction, EQ-5D-5L will be used to assess quality of life, and Pittsburgh Sleep Quality Index (PSQI) will be used to assess the quality of sleep. Data will be entered and analyzed through SPSS version 21.

DETAILED DESCRIPTION:
CABG Phase II rehabilitation typically begins a few weeks after hospital discharge and is a structured, medically supervised program aimed at stabilizing patients post-surgery. During this phase, patients often struggle with limited physical capacity, reduced exercise tolerance, and fatigue. Effective cardiac rehabilitation during this critical recovery phase is essential for optimizing health outcomes. Multimodal rehabilitation approaches have been shown to enhance recovery. The integration of innovative techniques like Virtual Reality (VR) into these multimodal programs can further engage patients. The objective of the study is to determine the effects of multimodal virtual reality-based rehabilitation on dyspnea, cardiorespiratory fitness, left ventricular ejection fraction, and quality of life in CABG phase II patients.

It will be a randomized clinical trial with a sample size of 66. A convenient sampling technique will be used to recruit the CABG phase II patients for the study. Then, they will be divided into three groups by block randomization. Weight-bearing Liuzijue Qigong will be given as a baseline treatment to all groups. In group A, patients will engage in multimodal circuit training while simultaneously viewing the nature scenes through VR in a clinical setting, in group B, patients will be given multimodal circuit training in a clinical setting while in group C, patients will be given multimodal circuit training through telerehabilitation. The dyspnea 12 Questionnaire will be used for measuring dyspnea, Cooper's 12-minute test will be used to assess cardiorespiratory fitness, echocardiography will be used to assess Left ventricular ejection fraction, EQ-5D-5L will be used to assess quality of life, and Pittsburgh Sleep Quality Index (PSQI) will be used to assess the quality of sleep. Data will be entered and analyzed through SPSS version 21.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent CABG surgery will be recruited after twelve weeks
* Both male and female
* Age 30-60 years old
* LVEF of < 40%
* Persistent dyspnea with a self-rated intensity of ⩾5 (out of 10) on a visual analogue dyspnea scale (this dyspnea rating was only used as an inclusion criterion and not as a measure for outcome)
* Preserved cognitive function (Montreal Cognitive Assessment score >24)

Exclusion Criteria:

* Patient with recurrent history of CABG
* Had a non-cardiac surgical procedure ≤2 months prior to recruitment
* Unstable angina, uncontrolled hypertension (blood pressure >180/100 mmHg), a pacemaker or atrial fibrillation, documented peak orifice area valve stenosis, symptomatic peripheral arterial disease that limits exercise capacity.
* Documented chronic obstructive pulmonary disease (FEV1 <60% and FVC <60%)
* Any shoulder impairment that would limit exercise participation
* Patients with Kinesiophobia
* Epilepsy, vertigo, eyesight impairment (conditions contraindicated for VR)

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
dyspnea by Dyspnea 12 questionnaire | 2 months
  This 12-item questionnaire was developed to measure the severity of dyspnea. The first seven items of this 4-point Likert-type scale (0 = none, 1 = mild, 2 = moderate, 3 = severe) ask patients about physical difficulties they experience because of dyspnea. The remaining five items of the questionnaire focus on the affective aspects of breathing. The maximum scores for the physical and affective aspects of the questionnaire are 21 and 15, respectively. The minimum total score for the questionnaire is 0, whereas the maximum total score is 36.The higher the score, the more severe will be the dyspnea.
cardiorespiratory fitness by VO2 max (through Cooper 12 min test) | 2 months
  Cooper proposed an indirect approach to estimate VO2 max based on field data. The test can be easily implemented in a common 400 m track field. After a warmup period of about 10 min, subjects are asked to run/ walk as much distance as possible for 12 min. Cooper conducted the test for 105 subjects and found a positive correlation with the value of VO2max quantified via a formal treadmill test. Cooper used linear regression of the covered distance versus the treadmill-estimated VO2 max to find the following relationship:
  VO 2 max ≈ 11.288+22.351D12.
left ventricular ejection fraction [LVEF] by echocardiography | 2 months
  LVEF (Left Ventricular Ejection Fraction) by echocardiography is a key measure of heart function, representing the percentage of blood pumped out of the left ventricle with each heartbeat. It is commonly used to assess cardiac efficiency and detect heart failure or other cardiovascular conditions. Echo provides a non-invasive, real-time evaluation of LVEF, offering insights into the heart's pumping capacity and overall health.
Quality of life by EQ-5D-5L | 2 months
  The EQ-5D questionnaire was developed to measure self-reported health simply and generically. It contains a descriptive system that includes the five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/ depression, and a visual analogue scale (the EQ VAS). Both the descriptive system and the EQ VAS measure the current health of the respondent. Combining the respondents' answers in each of the five dimensions of the descriptive system results in a unique health state. On the EQ-VAS, the respondents rate their current health on a scale ranging from 0 to 100. Zero represents "the worst health you can imagine" and 100 represents "the best health you can imagine".

SECONDARY OUTCOMES:
Sleep by Pittsburgh Sleep Quality Index (PSQI) | 2 months
  The PSQI is an 18-item constructed questionnaire designed to assess overall sleep quality over 1 month. The 18 items are divided into 7 derived component scores: (1) sleep quality, (2) sleep latency, (3) sleep duration, (4) sleep efficiency, (5) sleep disturbance, (6) medication use and (7) daytime dysfunction. These items are rated in terms of the frequency or severity of the problem on a four-point Likert scale (e.g., 0 = Not during the past month, 1 = Less than once a week, 2 = Once or twice a week, 3 = Three or more times a week). The sum of the component scores yields a global PSQI score that ranges from 0 to 21, with higher scores representing lower sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Wajeeha Zia, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

REFERENCES:
- [Background] Elbrond P, Hojskov IE, Missel M, Borregaard B. Food and heart-the nutritional jungle: Patients' experiences of dietary habits and nutritional counselling after coronary artery bypass grafting. J Clin Nurs. 2020 Jan;29(1-2):85-93. doi: 10.1111/jocn.15061. Epub 2019 Oct 2. PMID 31512796
- [Background] Ramos-Campo DJ, Andreu Caravaca L, Martinez-Rodriguez A, Rubio-Arias JA. Effects of Resistance Circuit-Based Training on Body Composition, Strength and Cardiorespiratory Fitness: A Systematic Review and Meta-Analysis. Biology (Basel). 2021 Apr 28;10(5):377. doi: 10.3390/biology10050377. PMID 33924785
- [Background] Zamzmi G, Rajaraman S, Hsu LY, Sachdev V, Antani S. Real-time echocardiography image analysis and quantification of cardiac indices. Med Image Anal. 2022 Aug;80:102438. doi: 10.1016/j.media.2022.102438. Epub 2022 Jun 9. PMID 35868819
- [Background] Gungor S, Tosun B, Unal N, Dusak I. Evaluation of dyspnea severity and sleep quality in patients with novel coronavirus. Int J Clin Pract. 2021 Oct;75(10):e14631. doi: 10.1111/ijcp.14631. Epub 2021 Jul 20. PMID 34260144
- [Background] Rutkowski S, Szczegielniak J, Szczepanska-Gieracha J. Evaluation of the Efficacy of Immersive Virtual Reality Therapy as a Method Supporting Pulmonary Rehabilitation: A Randomized Controlled Trial. J Clin Med. 2021 Jan 18;10(2):352. doi: 10.3390/jcm10020352. PMID 33477733
- [Background] Jozwik S, Cieslik B, Gajda R, Szczepanska-Gieracha J. Evaluation of the Impact of Virtual Reality-Enhanced Cardiac Rehabilitation on Depressive and Anxiety Symptoms in Patients with Coronary Artery Disease: A Randomised Controlled Trial. J Clin Med. 2021 May 16;10(10):2148. doi: 10.3390/jcm10102148. PMID 34065625
- [Background] Moneruzzaman M, Sun WZ, Changwe GJ, Wang YH. Efficacy of Multiple Exercise Therapy after Coronary Artery Bypass Graft: A Systematic Review of Randomized Control Trials. Rev Cardiovasc Med. 2023 May 9;24(5):141. doi: 10.31083/j.rcm2405141. eCollection 2023 May. PMID 39076757
- [Background] Dimitriadis S, Qian E, Irvine A, Harky A. Secondary Prevention Medications Post Coronary Artery Bypass Grafting Surgery-A Literature Review. J Cardiovasc Pharmacol Ther. 2021 Jul;26(4):310-320. doi: 10.1177/1074248420987445. Epub 2021 Jan 29. PMID 33514291
- [Background] Montrief T, Koyfman A, Long B. Coronary artery bypass graft surgery complications: A review for emergency clinicians. Am J Emerg Med. 2018 Dec;36(12):2289-2297. doi: 10.1016/j.ajem.2018.09.014. Epub 2018 Sep 8. PMID 30217621
- [Background] Pooria A, Pourya A, Gheini A. Postoperative complications associated with coronary artery bypass graft surgery and their therapeutic interventions. Future Cardiol. 2020 Sep;16(5):481-496. doi: 10.2217/fca-2019-0049. Epub 2020 Jun 4. PMID 32495650
- [Background] McNichols B, Spratt JR, George J, Rizzi S, Manning EW, Park K. Coronary Artery Bypass: Review of Surgical Techniques and Impact on Long-Term Revascularization Outcomes. Cardiol Ther. 2021 Jun;10(1):89-109. doi: 10.1007/s40119-021-00211-z. Epub 2021 Jan 30. PMID 33515370